CLINICAL TRIAL: NCT04462900
Title: Multi-center, Single Arm, Observational Study to Evaluate the Safety of Linaclotide in IBS-C Patients in China
Brief Title: Evaluate the Safety of Linaclotide in IBS-C Patients in China
Acronym: Liberty
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5630R00001
Record Dates: First submitted 2020-06-19; First posted 2020-07-08 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-03

CONDITIONS: Irritable Bowel Syndrome-IBS
Keywords: IBS
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: None Retained — no sample collect in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a Multi-center, single arm, observational study to evaluate the safety of linaclotide in IBS-C patients in China. Enrolls approximately 3,000 Chinese patients from 30 participating sites around China and followed up for half year.

DETAILED DESCRIPTION:
This is a multi-center, one arm, prospective observational study which enrolls approximately 3,000 Chinese patients in China.The study will be performed under real world clinical practice setting. Patients will be eligible for the study after taking at least one dose of linaclotide. Every patient will be followed maximum of 6 months after enrollment. Study measures will be collected at baseline and during the follow-up period. Incidence of adverse events will be employed to assess the safety and tolerability of linaclotide in Chinese patients. The treatment satisfaction will be employed to assess the impact of treatment. The Irritable Bowel Syndrome-Quality of Life Measure (IBS-QoL) will be employed to assess the patient's quality of life.

ELIGIBILITY:
Inclusion Criteria:

* ≧ 18 years old
* Provision of subject informed consent prior to any study procedures
* Has taken at least one dose of linaclotide
* NOT participating in any interventional study currently or during the last 3 months

Exclusion Criteria:

* If linaclotide is contraindicated according to the product prescribing information
* Being unable to comply with study-specified procedure
* Has ever participated in current study before -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 3,000 Chinese patients in China, Patients will be eligible for the study after taking at least one dose of linaclotide. Duration will from 2020 Q2 to 2023 Q1.
Sampling Method: Probability Sample
Enrollment: 3028 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Demonstrate the safety of linaclotide therapy | 2023/09/30
  The primary objective of current study is to demonstrate the safety of linaclotide therapy by assessment of the incidence of any adverse events (AEs) , serious adverse events (SAEs) , AEs by severity, ADRs and AEs leading to linaclotide-associated interruption, discontinuation, and death during 6-month follow up in Chinese patients.

SECONDARY OUTCOMES:
Assess the treatment satisfaction | 2023/09/30
  To observe patients' treatment satisfaction status after treatment via a 5-point treatment satisfaction scale (1=not at all, 2=a little, 3=somewhat, 4=very, 5=extremely)
Assess the impact of linaclotide treatment in patient's quality of life. | 2023/09/30
  To describe patient's quality of life after treatment via the Irritable Bowel Syndrome-Quality of Life Measure (IBS-QoL).

CONTACTS AND LOCATIONS:
Locations (22):
- China (22):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Binzhou
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Jinan
  - Research Site, Leshan
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Suzhou
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Ürümqi
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Zhengzhou

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5630R00001&attachmentIdentifier=7476fb16-53fe-40bc-aef7-6b9849920507&fileName=AZ_liberty_CSR_synopsis.pdf&versionIdentifier=